CLINICAL TRIAL: NCT07046260
Title: Prospective Cohort Study With Case Enrichment to Assess a Diagnostic Aid for Cancer in Symptomatic Subjects (PROCARES)
Brief Title: Prospective Study to Assess a Diagnostic Aid for Cancer
Acronym: PROCARES
Status: Recruiting | Type: Observational
Sponsor: Harbinger Health (Industry)
Responsible Party: Sponsor
Other Study IDs: HH-PRT-0005
Record Dates: First submitted 2025-06-09; First posted 2025-07-01 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-08

CONDITIONS: Cancer
Keywords: Cancer; Diagnostic; Oncology; Test; Observational
MeSH Terms: conditions — Neoplasms; Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with clinical suspicion of cancer or patients recently diagnosed with Cancer: People who have signs, symptoms, and/or findings that their doctor suspects may be related to cancer, or who have recently been diagnosed with cancer and have not received treatment for this cancer.
  Interventions: Other: Blood sample collection

INTERVENTIONS:
Other: Blood sample collection — The study will collect up to 40 mL of whole peripheral blood in Streck Cell-Free DNA BCT® tubes from each Subject.
  Other Names: Diagnostic Aid Test

SUMMARY:
The primary objective of this study is to evaluate the performance of a blood-based diagnostic aid test for cancer detection in individuals presenting with symptoms, signs, or findings that raise clinical suspicion for cancer.

DETAILED DESCRIPTION:
Subjects 45 years of age and older presenting with symptoms, signs, and/or findings suggestive of one or more cancers originating from protocol-specified sites will be enrolled. Subjects will complete a blood draw for analysis by the investigational diagnostic aid test. For subjects with suspected cancer at enrollment, clinical outcomes will be determined following completion of a standard-of-care diagnostic work-up as clinically indicated. Subjects with a confirmed cancer diagnosis at enrollment must be treatment-naïve and will have diagnosis details collected at the time of enrollment. The results of the investigational diagnostic aid test will not be provided to investigators, treating clinicians, or subjects. Personnel performing clinical evaluations, determining final diagnoses, or reviewing diagnostic imaging and pathology reports will remain blinded to the results of the investigational test. All testing and associated analyses will be conducted in a blinded fashion, and test results will not inform clinical decision-making.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged ≥45 years at the time of informed consent
2. Provided written or electronic informed consent, according to local guidelines, signed and dated by the Subject or by a legal guardian prior to the performance of any study- specific procedures, sampling, or analyses
3. Presentation with symptoms, signs, and/or findings that raise clinical suspicion of one or more of the protocol-specified sites AND

   1. undergoing diagnostic work-up to determine if cancer is present, but do not yet have a confirmed cancer diagnosis. Subject must be willing to undergo a standard diagnostic work-up per local SoC to establish clinical truth regarding the presence or absence of cancer OR
   2. have a confirmed diagnosis of cancer, determined within 45 days prior to signing the Informed Consent Form, based on standard diagnostic procedures (histopathology, imaging, etc.) following presentation with symptoms, signs, and/or findings that raised a clinical suspicion of one or more cancers originating from the protocol-specified sites. Must be treatment-naïve for the diagnosed cancer at the time of enrollment.

Exclusion Criteria:

1. History of any prior invasive or hematological malignancy (Individuals with completely resected ductal carcinoma in-situ or non-melanoma skin cancer are permitted)
2. Subject is suffering from any febrile illness defined as a temperature >101.5°F within the last 48 hours
3. Subject is pregnant (Self-reported)
4. Subject is a recipient of an organ transplant, blood transfusion within 120 days, or prior non-autologous (allogeneic) bone marrow or stem cell transplant (Subject with a corneal transplant can be considered for study entry)
5. Inability or unwillingness to comply with study procedures or follow-up requirement
6. Previous or current participation in any study sponsored by, or employment with, Harbinger Health
7. Participation in a clinical research study sponsored by an external organization which may interfere with study procedures or outcomes
8. Subject has any condition that in the opinion of the Investigator should preclude participation in the study

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll individuals 45 years of age or older who present with symptoms, signs, and/or have findings leading to a clinical suspicion or a diagnosis of one or more cancers originating from the following sites:
  * Biliary Tract
  * Colon
  * Esophagogastric Junction (EGJ)
  * Esophagus
  * Gallbladder
  * Head and Neck
  * Liver
  * Lung
  * Lymphatic System
  * Ovary
  * Pancreas
  * Rectum
  * Stomach
Sampling Method: Non-Probability Sample
Enrollment: 1650 (Estimated)
Dates: Start 2025-07-11 (Actual); Primary Completion 2027-01-08 (Estimated); Study Completion 2027-05-25 (Estimated)

PRIMARY OUTCOMES:
Performance of a diagnostic aid test among individuals presenting with symptoms, signs, and/or clinical findings suggestive of one or more cancers originating from the protocol-specified sites. | 18 months
  * Proportion of positive test results among all confirmed cancer cases.
  * Proportion of negative test results among all subjects without a confirmed cancer diagnosis.
  * Proportion of subjects without a confirmed cancer diagnosis among all those who test negative.

SECONDARY OUTCOMES:
Intrinsic accuracy of the test separately within cancer types and stages. | 18 months
  * Sensitivity for early-stage (I and II) and late-stage (III and IV) cancer cases.
  * Sensitivity per cancer indication.
Effect of demographic covariates on the diagnostic performance of the test. | 18 months
  Performance metrics within clinically relevant subgroups defined by demographic factors.

CONTACTS AND LOCATIONS:
Overall Officials: Luke Pike, MD, DPhil, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (34):
- United States (34):
  - Palomar Health, Poway, California
  - Rocky Mountain Gastroenterology, Centennial, Colorado
  - Zoyla Almeida, MD PA, Coconut Creek, Florida
  - Azzi ENT and Facial Reconstructive Surgery, Jupiter, Florida
  - Prophase, LLC, Margate, Florida
  - Millennium Medical Research, Miami, Florida
  - Regis Clinical Research, Miami, Florida
  - Gastroenterology of Greater Orlando, Orange City, Florida
  - Millennium Physician Group, Port Charlotte, Florida
  - Stuart Oncology Associates, Stuart, Florida
  - Avita Clinical Research, Tampa, Florida
  - Pulmonary & Sleep Specialists of Northeast Georgia, P.C, Winder, Georgia
  - Christie Clinic, Champaign, Illinois
  - Hope and Healing Cancer Services, Hinsdale, Illinois
  - Iowa Clinic, West Des Moines, Iowa
  - Hutchinson Clinic, Hutchinson, Kansas
  - Northlake Gastroenterology Associates, Hammond, Louisiana
  - Velocity Clinical Research, Annapolis, Maryland
  - Capital Digestive Care, Chevy Chase, Maryland
  - Huron Gastroenterology, Ypsilanti, Michigan
  - Oncology Hematology Specialists, Mountain Lakes, New Jersey
  - Southwest Gastroenterology, Albuquerque, New Mexico
  - Westchester Putnam Gastro, Carmel, New York
  - Associated Gastroenterologists of Central New York, Fayetteville, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Wilmington Health, PLLC, Wilmington, North Carolina
  - Hightower Clinical, Oklahoma City, Oklahoma
  - Susquehanna Research Group, Harrisburg, Pennsylvania
  - Respiratory Specialists, Wyomissing, Pennsylvania
  - GIA Clinical Trials, LLC, Knoxville, Tennessee
  - Premier Family Physicians, Austin, Texas
  - Activian Clinical Research (Scarsdale), Houston, Texas
  - Huntsville Research Institute, LLC, Huntsville, Texas
  - Activian Clinical Research, Kingwood, Texas

IPD SHARING:
Plan to Share IPD: Undecided